CLINICAL TRIAL: NCT00311675
Title: A Single Center, Open-Label, Phase I/II Study of Two 90-µg Doses of Intramuscular Inactivated Influenza A/H5N1 Vaccine in Healthy Adult Subjects
Brief Title: St. Jude Open Label H5 Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-0130
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-07

CONDITIONS: Influenza
Keywords: influenza, A/H5N1, vaccine
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)

INTERVENTIONS:
Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur) — Monovalent subvirion H5N1 vaccine (HA of A/Vietnam/1203/04) provided in single-dose vials containing 90-mcg/mL A/H5N1 HA. Dosage is two 90 mcg doses administered intramuscularly separated by approximately 28 days.

SUMMARY:
The purpose of this study is to see how antibodies (proteins that fight infection) are made after you receive the new H5N1 flu vaccine. The new H5N1 vaccine will be given to 50 healthy adult lab workers, aged 18 years and older. Subjects will receive two 90mcg injections (shots in the arm) of the vaccine about 1 month apart. Subjects will maintain a memory aid to record oral temperature and any response to the vaccine for 7 days after each immunization. Subjects will be contacted by telephone 1 to 3 days after vaccination. They will return to the clinic on Day 7. Blood will be drawn before each vaccination and on Days 56 and 180. Subjects may be involved in the study for about 6 months. It is anticipated that the vaccine will provide safe protection against influenza H5N1.

DETAILED DESCRIPTION:
The purpose of this open-label, phase I/II study is to investigate the safety and immunogenicity of two 90-mcg doses of intramuscular inactivated influenza A/H5N1 vaccine in healthy adults, aged 18 years and older. Subjects will receive 2 doses of the vaccine separated by approximately 28 days. Subjects will maintain a memory aid to record oral temperature and systemic and local adverse events (AEs) for 7 days after each immunization. Subjects will be contacted by telephone 1 to 3 days after vaccination (approximately Day 2) to assess concomitant medications and the occurrence of AEs, and they will return to the clinic on Day 7 for AE and concomitant medication assessment, a targeted physical examination (if indicated), and review of the memory aid. Serum for immunogenicity evaluations will be obtained prior to the first vaccination (Day 0) and prior to the second vaccination (at Day 28), and on Days 56 and 180. Primary objectives are to determine the safety of subvirion inactivated A/H5N1 vaccine in healthy adults and to determine the immunogenicity of subvirion inactivated H5N1 vaccine in healthy adults approximately 1 month following receipt of each of two 90 mcg doses of vaccine. The secondary objective is to evaluate immunogenicity and the percent of subjects responding approximately 1 and 7 months after the first vaccination. Primary endpoints are: AE or serious adverse event information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessment); geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers 28 days after receipt of second dose of the vaccine; and GMT and frequency of 4-fold or greater increases in serum hemagglutination inhibition (HAI) antibody titers against the influenza A/H5N1 virus 28 days after receipt of the second dose of the vaccine. The secondary endpoints are GMT and frequency of 4-fold or greater increases in neutralizing antibody titers in each group 1 month and 7 months after receipt of the first dose of vaccine; GMT and frequency of 4-fold or greater increases in serum hemagglutination inhibition (HAI) antibody titers in each group 1 month and 7 months after receipt of the first dose of vaccine; and development of serum antibody responses against antigenically drifted variants of H5N1 influenza viruses.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory personal with potential exposure to live H5N1 viruses.
* Male or nonpregnant female (as indicated by a negative urine pregnancy test prior to each dose of vaccine), aged 18 years and older.
* Women of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (i.e., barrier method, abstinence, and licensed hormonal methods) for the entire study period.
* Is in good health, as determined by vital signs (pulse, blood pressure, oral temperature), medical history, and a targeted physical examination based on medical history.
* Able to understand and comply with planned study procedures.
* Provides informed consent prior to any study procedures and is available for all study visits.

Exclusion Criteria:

* Has a known allergy to eggs or other components of the vaccine.
* Has a known allergy or sensitivity to latex (in the stopper).
* Has a positive urine pregnancy test prior to vaccination (if female of childbearing potential) or women who are breastfeeding.
* Is undergoing immunosuppression as a result of an underlying illness or treatment.
* Has an active neoplastic disease or a history of any hematologic malignancy.
* Is using oral or parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs.
* Has a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Has an acute illness, including an oral temperature greater than 100.4 degrees F, within 1 week of vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during the 6-month study period.
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Adverse event (AE) or serious AE information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessment). | 1 - 3 days after each vaccination to review any AEs and SAEs; approximately 1 week after each vaccination review any AEs and collect for 28 days following the 2nd dose of vaccine. SAEs will be collected throughout the study through day 180.
Geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers. | 28 days after receipt of 2nd dose of vaccine.
Geometric mean titer (GMT) and frequency of 4-fold or greater increases in serum hemagglutination inhibition (HAI) antibody titers against the influenza A/H5N1 virus. | 28 days after receipt of 2nd dose of vaccine.

SECONDARY OUTCOMES:
Geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers in each group. | 1 month and 7 months after receipt of the first dose of vaccine.
Geometric mean titer (GMT) and frequency of 4-fold or greater increases in serum hemagglutination inhibition (HAI) antibody titers in each group. | 1 month and 7 months after receipt of the first dose of vaccine.
Development of serum antibody responses against antigenically drifted variants of H5N1 influenza viruses. | Serum for immunogenicity evaluations will be obtained prior to the 1st vaccination (day 0) and prior to the 2nd vaccination (day 28), and on days 56 and 180.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States